CLINICAL TRIAL: NCT06436638
Title: Comparison of Nasal Continuous Positive Airway Pressure (CPAP) Mask and Nasal Airway in Terms of Intraoperative Anesthesia Quality and Postoperative Associated Complications in Impacted Molar Tooth Extraction Patients Under Deep Sedation; A Multi-Center Study
Brief Title: Comparison of Nasal Continuous Positive Airway Pressure (CPAP) Mask and Nasal Airway in Molar Tooth Extraction Under Deep Sedation
Status: Recruiting | Type: Observational
Sponsor: Gözde Nur Erkan (Other)
Collaborators: TC Erciyes University (Other); Kırıkkale University (Other)
Responsible Party: Sponsor-Investigator, Gözde Nur Erkan, Assistant Professor Doctor, Medical Doctor, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: KU-ERKAN-001
Record Dates: First submitted 2024-05-10; First posted 2024-05-31 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Deep Sedation; Non-invasive Ventilation Support; Nasal Airway; Nasal CPAP Mask; Impacted Molar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Airway: Group to receive non-invasive ventilation support via nasal airway during dental extraction under deep sedation.
  Interventions: Device: Non-invasive ventilation support equipment
- Group Mask: Group to receive non-invasive ventilation support via nasal CPAP mask during dental extraction under deep sedation
  Interventions: Device: Non-invasive ventilation support equipment

INTERVENTIONS:
Device: Non-invasive ventilation support equipment — Non-invasive ventilation support is provided by nasal airway and nasal CPAP mask to avoid respiratory complications such as hypoxia, desaturation, hypercarbia, respiratory depression etc. during extraction of impacted molars under deep sedation.

SUMMARY:
In patients with high levels of fear and anxiety, it is recommended to perform dental procedures under sedation or general anesthesia depending on the nature of the procedure. In dental treatment under anesthesia, it is important that the procedure is comfortable and well tolerated by the patient. In addition, patient comfort is important in all dental procedures to prevent the development of avoidance behavior.

During dental procedures performed under anesthesia, the oral cavity is completely within the scope of the surgical or procedure field. In this respect, sedation and general anesthesia in dental procedures and operations have specific risks and challenges.Since there is a risk of respiratory depression, hypoxia and hypercarbia during deep sedation, non-invasive ventilation support provided to patients with airway devices would be beneficial. In the research clinics where the study will be conducted, deep sedation with non-invasive mechanical ventilation support using a nasal CPAP (Continuous Positive Airway Pressure) mask or nasal airway is applied during the extraction of impacted molars. Thus, many dental procedures are routinely performed under deep sedation without the need for general anesthesia. There are very limited data in the literature on the use of a nasal CPAP mask during sedation for different procedures in patients with obstructive sleep apnea or obesity. However, no study comparing ventilation support during deep sedation with nasal CPAP mask and nasal airway has been found in the literature.

The aim of this study is to compare the non-invasive ventilation support provided with 2 different airway devices during the procedure in terms of intraoperative and postoperative related complications, ventilation parameters, patient and surgeon satisfaction.

The hypothesis of the study is that two different ventilation support methods during deep sedation may be superior to each other in terms of anesthesia quality, postoperative complications related to airway devices, patient and surgeon satisfaction.

In the study, a total of 60 patients (Group airway, n;30, Group Mask, n;30) from 2 centers are planned to be included in the study by performing power analysis with a statistical power of the trial >0.8.

The permutation method will be applied within the scope of the restricted randomization method to determine the group of patients to be included.

DETAILED DESCRIPTION:
In the study to be conducted in two dental faculties, it is planned to use a total of 60 patient data, 30 patients with nasal CPAP mask and 30 patients with nasal airway. In the centers where the study will be conducted, deep sedation during dental procedures with ventilatory support via nasal airway and nasal CPAP mask, which will be compared in the study, is applied in routine practice. In this context, anxiolysis with 2 mg IV midazolam is administered to the patients before they are taken to the operating room on the day of the procedure. Patients are administered 1.5 mg/kg propofol and 0.5 mcg/kg fentanyl intravenously for sedation induction. Non-invasive ventilation support is then applied with a nasal airway or nasal CPAP mask and ventilation parameters are screened. Sevoflurane at 1 MAC (minimum alveolar concentration) level is administered inhalationally for sedation maintenance and the level of sedation is evaluated using the Ramsey sedation scale. Surgical dental extraction procedures between 20-60 minutes will be included in the study. For postoperative analgesia, paracetamol 1 g and dexketoprofen trometamol 50 mg are administered intravenously. The data planned to be collected within the scope of the study are blood pressure, heart rate, peripheral oxygen saturation (number of desaturation episodes), respiratory rate, ventilation parameters (Tidal volume (TV); set and actual, minute volume , end tidal CO2-EtCO2, and Peak pressure (Peak P). The total dose of agents used for sedation will also be recorded. During the post-operative follow-up period, the presence of nausea-vomiting, nasal pain, dryness in the nasal mucosa, epistaxis, sore throat, and dryness in the throat will be evaluated. Patient and surgeon satisfaction scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer adult patients aged 18-60 years
* Patients scheduled for impacted tooth extraction
* Cases with surgical time ≥20 minutes and ≤60 minutes
* American Society of Anaesthesiologists (ASA) physical status I and II patients
* Patients with BMI≤30

Exclusion Criteria:

* Patients under 18 years old-over 60 years old
* Surgeries with a procedure time over 1 hour or less than 20 minutes
* American Society of Anaesthesiologists (ASA) physical status III and higher patients
* Presence of conditions such as mental retardation that impair the patient's ability to make decisions about himself/herself
* Patients with respiratory system diseases such as asthma, chronic obstructive pulmonary disease (COPD) or airway hyperreactivity
* Patients with a condition that severely narrows the nasal passage opening (e.g. adenoid hypertrophy, etc.)
* Patients with BMI>30
* Patients who refused to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: It is planned to investigate patients with a diagnosis of impacted molars, who have an indication for dental extraction, and who are scheduled for dental extraction under sedation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Non-invasive blood pressure | Intraoperative period and for 4 hours after surgery
  It is planned to record non-invasive blood pressure values of the patients at regular intervals during the operation, recovery unit and inpatient ward follow-up. Changes in blood pressure above 20% from baseline will be recorded additionally.
ECG | Intraoperative period and for 4 hours after surgery
  It is planned to record heart rate values of the patients at regular intervals during the operation, recovery unit and inpatient ward follow-up. Changes in heart rate greater than 20% of baseline will be recorded additionally.
Peripheral oxygen saturation | Intraoperative period and for 4 hours after surgery
  It is planned to record peripheral oxygen saturation values of the patients at regular intervals during the operation, recovery unit and inpatient ward follow-up. Hypoxia (SpO2<90%) will be recorded additionally.
Respiratory rate | Intraoperative period and for 4 hours after surgery
  It is planned to record respiratory rate values of the patients at regular intervals during the operation, recovery unit and inpatient ward follow-up. Respiratory depression will be recorded additionally.
Number of interruptions for an anesthesia-related reason | Intraoperative period
  Number of episodes during deep sedation when the procedure has to be interrupted due to desaturation or patient movement will be recorded
Tidal volume | Intraoperative period
  During non-invasive ventilatory support, set and actual tidal volume values will be recorded at regular intervals during the operation.
Peak pressure | Intraoperative period
  During non-invasive ventilatory support, peak pressure values will be recorded at regular intervals during the operation.
End tidal carbon dioxide level (EtCO2) | Intraoperative period
  During non-invasive ventilatory support, end tidal carbon dioxide values will be recorded at regular intervals during the operation.
Minute ventilation | Intraoperative period
  During non-invasive ventilatory support, minute ventilation values will be recorded.

SECONDARY OUTCOMES:
Postoperative complications related non-invasive ventilation support devices and sedation | During the next 3 hours after the end of the operation
  During the recovery unit and inpatient ward follow-up, patients will be monitored for the presence of nausea/vomiting, pain and/or itching/dryness in the nose and/or throat. A 10-point Likert scale would be used for nausea and vomiting assessment (0 points: No nausea, 1-2 points: Very mild nausea, 3-4 points: Mild nausea, 5-6 points: Moderate nausea, 7-8 points: Severe nausea and 9-10 points: worst nausea). For pain, a 10-point visual analog scale would be used. Additionally, the development of epistaxis will be recorded.
Patient and surgeon satisfaction | Perioperative period
  Using a 5-point Likert scale, the satisfaction level of the patients and the surgeon will be questioned and recorded. In the Likert scale, 5 indicates the highest level of satisfaction and 1 indicates the lowest level of satisfaction.
Total dose of medications used for sedation during the procedure | Intraoperative period
  The total dose of anesthetic medications required to provide a depth of sedation with a Ramsey sedation score of 5 or higher during the surgical procedure will be recorded
Recovery duration from anesthesia | From the end of the operation until discharge to the ward
  The time until the Modified Aldrete Score is 9 or higher during the recovery period

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University Faculty of Dentistry, Kayseri
  - Kırıkkale University Faculty of Dentistry, Kırıkkale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appukuttan DP. Strategies to manage patients with dental anxiety and dental phobia: literature review. Clin Cosmet Investig Dent. 2016 Mar 10;8:35-50. doi: 10.2147/CCIDE.S63626. eCollection 2016. PMID 27022303
- [Background] Cukierman DS, Perez M, Guerra-Londono JJ, Carlson R, Hagan K, Ghebremichael S, Hagberg C, Ge PS, Raju GS, Rhim A, Cata JP. Nasal continuous positive pressure versus simple face mask oxygenation for adult obese and obstructive sleep apnea patients undergoing colonoscopy under propofol-based general anesthesia without tracheal intubation: A randomized controlled trial. J Clin Anesth. 2023 Oct;89:111196. doi: 10.1016/j.jclinane.2023.111196. Epub 2023 Jul 3. PMID 37406462
- [Background] Bai Y, Xu Z, Chandrashekar M, St Jacques PJ, Liang Y, Jiang Y, Kla K. Comparison of a simplified nasal continuous positive airways pressure device with nasal cannula in obese patients undergoing colonoscopy during deep sedation: A randomised clinical trial. Eur J Anaesthesiol. 2019 Sep;36(9):633-640. doi: 10.1097/EJA.0000000000001052. PMID 31313720